CLINICAL TRIAL: NCT01537003
Title: WOUNDCHEK™ Protease Status Point of Care (POC) Diagnostic Test A Prospective, Multi Centre, Randomised, Clinical Study on Venous Leg Ulcers
Brief Title: WOUNDCHEK™ Protease Status Point of Care (POC) Diagnostic Test
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Systagenix Wound Management (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SWM1200
Record Dates: First submitted 2012-02-16; First posted 2012-02-22 (Estimated); Last update posted 2013-07-08 (Estimated); Status verified 2013-05

CONDITIONS: Venus Leg Ulcers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Promogran and Low EPA (Experimental): Patients with low EPA will be treated with PROMOGRAN and standard of care for vlu compression
  Interventions: Device: Promogran
- Low EPA and compression (Active Comparator): Patients with Low EPA will only get standard of care for VLU which is compression.
  Interventions: Device: Coban 2 layer
- High EPA and compression (Active Comparator): Patients with high EPA will get standard of care for VLU which is compression.
  Interventions: Device: Coban 2 layer
- Promogran High EPA (Experimental): patients with HIGH EPA will then be treated with PROMOGRAN and standard of care for VLU compression
  Interventions: Device: Promogran

INTERVENTIONS:
Device: Promogran — Promogran is a collagen/ORC dressing which modulates the wound environment
  Arms: Promogran High EPA; Promogran and Low EPA
Device: Coban 2 layer — Compression bandage
  Arms: High EPA and compression; Low EPA and compression

SUMMARY:
The purpose of this trial is to determine if wounds with elevated protease activity (EPA) treated with targeted interventions such as protease modulating therapies can improve clinical and economic outcomes.

Multi-centre VLU study to investigate efficacy of WOUNDCHEK™ on EPA wounds

DETAILED DESCRIPTION:
The purpose of this trial is to determine if wounds with elevated protease activity (EPA) treated with targeted interventions such as protease modulating therapies can improve clinical and economic outcomes. It is hypothesized that protease modulating dressings may provide significantly better clinical outcomes on EPA wounds over current standard of care.

Wounds with EPA will be determined using a new POC diagnostic test, WOUNDCHEK™ Protease Status, and the efficacy of PROMOGRAN®, a protease modulating therapy will be determined against standard of care (moist wound healing and compression) in VLU wounds in both elevated EPA and low protease activity wounds.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged ≥ 18 years old
* Patients with a leg ulcers of venous aetiology as determined by ankle brachial pressure index (ABPI) ≥ 0.8 and able and willing to use appropriate compression therapy
* Duration of ulcer ≥ 6 weeks ≤ 3 years
* Ulcer is ≥ 1 cm2 ≤ 100cm2 no length longer than 10cm
* The patient must be able to understand the trial and provide written informed consent
* No local or systemic signs of infection, with normal CRP and leukocyte levels below 10 000
* Wound has not been treated with PROMOGRAN® in 4 weeks prior to inclusion

Exclusion Criteria:

* Leg ulcers that do not have venous aetiology as determined by not been suitable for compression therapy and having an ABPI ≤ 0.8
* Leg ulcer smaller than 1cm2 and larger than 100cm2 and has any length longer than 10cm
* Wound duration of less than 6 weeks or longer than 3 years
* Known hypersensitivity to any of the wound dressing used in the trial
* Current local or systemic antibiotics in the week prior to inclusion
* Clinical infected wound as determined by the presence of 3 or more of the following clinical signs: perilesional erythema, pain between two dressing changes, malodorous wound, abundant exudate and oedema.
* Progressive neoplastic lesion treated by radiotherapy or chemotherapy
* Prolonged treatment with immunosuppressive agents or high dose corticosteroids
* Patients who have a current illness or condition which may interfere with wound healing in the last 30 days (carcinoma, connective tissue disease, autoimmune disease or alcohol or drug abuse)
* Life expectancy of <6 months
* Patients with uncontrolled diabetes as determined by Hb-A1c ≥ 12% ( = Hb-1CIFCC ≥ 107.65 mmol/mol)
* Patients who have participated in a clinical trial on wound healing within the past month
* Patients who are unable to understand the aims and objectives of the trial
* Patients with a known history of non adherence with medical treatment
* Females who are pregnant
* Subject has Acquired Immunodeficiency Syndrome (AIDS) or is known to be infected with Human Immunodeficiency Virus (HIV)
* Subject has viral hepatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-10 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
The primary end-point of this study will be to identify EPA wounds using WOUNDCHEK™ Protease Status diagnostic test | 12 weeks
  The primary end-point of this study will be to identify EPA wounds using WOUNDCHEK™ Protease Status diagnostic test, and to compare the healing outcomes of two treatment regimes (PROMOGRAN®, a protease modulating therapy and current standard of care) on chronic wounds with EPA.
  An improved healing outcome for venous leg ulcers will be defined as the proportion of wounds which reach a minimum 30% percentage reduction in wound surface area over a four-week treatment period.

SECONDARY OUTCOMES:
The average percentage change in protease activity levels pre and post treatment | 12 weeks
  The proportion of wounds achieving wound closure (defined as a restoration of a complete epithelial cover) at twelve weeks and the average time to wound closure. The relative cost effectiveness of both treatment regimes when they are targeted appropriately; PROMOGRAN®, a protease modulating therapy targeted to wounds with EPA and standard of care to wounds with LPA.Healing outcomes for standard of care on EPA wounds as compared to LPA wounds.
  Healing outcomes for PROMOGRAN®, a protease modulating therapy on EPA wounds as compared to LPA wounds.

CONTACTS AND LOCATIONS:
Overall Officials: Keith Harding, Prof, Principal Investigator — Cardiff University
Locations (7):
- Penn North Centers for Advance Wound Care, Eire, Pennsylvania, United States
- Germany (2):
  - University Medical Center Gieben and Marburg GmBH, Marburg
  - Dres. Bolko Alter Siamak Pourhassan, Oberhausen
- Italy (2):
  - University of Pisa, Pisa, Roma
  - University of Ferrara, Ferrara
- United Kingdom (2):
  - Cardiff University, Cardiff, Wales
  - Bradford Royal Infirmary, Bradford, Yorkshire